CLINICAL TRIAL: NCT04596371
Title: A Single-center Prospective Cohort Study for Pure Pulmonary Ground Glass Nodules in Women Preparing for Pregnancy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: B2019-335
Record Dates: First submitted 2020-10-11; First posted 2020-10-22 (Actual); Last update posted 2020-10-22 (Actual); Status verified 2020-01

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms | interventions — Pregnancy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: pure pulmonary ground glass nodules in women preparing for pregnancy — pure pulmonary ground glass nodules in women preparing for pregnancy

SUMMARY:
In this study, about 200 pure GGO in women preparing for pregnancy will be included for a 5-year follow-up. The aim of this study is to elucidate the biological nature of pulmonary GGO lesion in women preparing for pregnancy and provide evidence for GGO treatment.

ELIGIBILITY:
Inclusion Criteria:

- 20-45 years' old found pulmonary GGO with chest CT scan and CT follow-up after 3 months shows that the GGO remains Diameter of GGO > 5mm and < 3cm

Exclusion Criteria:

- receiving immunosuppressor or steriods receiving chemo- or radio- therapy can not receive regular follow-up

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: pure pulmonary ground glass nodules in women preparing for pregnancy
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2020-11-01 (Estimated); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes from baseline GGO diameter | 6 months, 1year, 2 years, 3 years, 4 years and 5 years
  Changes from baseline GGO diameter
Changes from baseline GGO CT index. | 6 months, 1year, 2 years, 3 years, 4 years and 5 years
  Changes from baseline GGO CT index.

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongshan Hospital, Shanghai, Shanghai Municipality, China